CLINICAL TRIAL: NCT05271058
Title: Effect of Intracameral Steroids Injection During Phacoemulsification on Postoperative Corneal Edema and Corneal Endothelium
Brief Title: Effect of Intracameral Steroids During Phacoemulsification on the Cornea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, khaled gamal abueleinen, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMBSUREC/30042019/Mohamed
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Corneal Edema
MeSH Terms: conditions — Corneal Edema | interventions — Control Groups; Triamcinolone; Population Groups

STUDY DESIGN:
Intervention Model Description: Purpose: Investigating the effect of intracameral steroids at the end of phacoemulsification on corneal edema and endothelial count.
  Methods: Prospective, interventional case control study. Sixty-nine eyes were randomized into 3 groups, 23 eyes each : 2groups received intracameral dexamethasone and triamcinolone (TA) respectively, while controls didn't receive any intraoperative steroids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group 1 (Sham Comparator): 23 eyes that did not receive any intraoperative steroids
  Interventions: Other: Control group
- Dexamethasone group 2 (Active Comparator): 23 eyes that received intracameral dexamethasone
  Interventions: Drug: Dexamethasone group
- Triamcinolone (TA) group 3 (Active Comparator): 23 eyes that received intracameral triamcinolone (TA)
  Interventions: Drug: Triamcinolone (TA) group

INTERVENTIONS:
Other: Control group — 23 eyes that didn't receive any intraoperative steroids
  Other Names: No intraoperative steroids
  Arms: Control group 1
Drug: Dexamethasone group — 23 eyes each received intracameral dexamethasone at the conclusion of phacoemulsification Received intracameral 0.4 mg in / 0.1 ml dexamethasone (8mg/2ml®; Amriya or Epico) at the end of phacoemulsification.
  Other Names: Intracameral Dexamethasone
  Arms: Dexamethasone group 2
Drug: Triamcinolone (TA) group — 23 eyes each received intracameral triamcinolone (TA) at the conclusion of phacoemulsification Received intracameral 2 mg/0.05 ml triamcinolone (TA) (Kenacort-A®; Bristol-Myers Squibb) at the end of phacoemulsification.
  Other Names: Intracameral triamcinolone (TA)
  Arms: Triamcinolone (TA) group 3

SUMMARY:
Prospective, interventional case control study. Sixty-nine eyes were randomized into 3 groups, 23 eyes each : 2groups received intracameral dexamethasone and triamcinolone (TA) respectively, while controls didn't receive any intraoperative steroids.

Intracameral steroids at the conclusion of phacoemulsification significantly improved corneal edema and spared corneal endothelium.

DETAILED DESCRIPTION:
Purpose: Investigating the effect of intracameral steroids at the end of phacoemulsification on corneal edema and endothelial count.

Methods: Prospective, interventional case control study. Sixty-nine eyes were randomized into 3 groups, 23 eyes each : 2groups received intracameral dexamethasone and triamcinolone (TA) respectively, while controls didn't receive any intraoperative steroids.

On the first postoperative day corneal edema in control compared to dexamethasone and TA groups respectively.

One month later, the mean increase of corneal thickness in control compared to intracameral dexamethasone and TA groups, respectively.

mean endothelial cell loss in control compared to intracameral dexamethasone and TA groups respectively.

ELIGIBILITY:
Inclusion Criteria:

* Cataract grades 2 to 5 nuclear cataract (LOCS III scale)
* uneventful phacoemulsification operation

Exclusion Criteria:

* extremely hard cataract grade 6 nuclear cataract (LOCS III scale)
* soft cataract
* subluxated lenses or zonular dehiscence
* associated ocular pathology such as glaucoma
* any signs of uveitis
* trauma
* retinal detachment
* vitrectomized or silicone filled eyes
* corneal disease such as Fuch's dystrophy, corneal opacity
* previous refractive corneal surgery
* Cases that developed ruptured posterior capsule and vitreous loss
* those lost to follow up were excluded and randomly replaced by the next chronological patient

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Corneal edema | First day postoperative
  Clinical grade of corneal edema on the first postoperative day
Central corneal thickness (CCT) | Three months
  Central corneal thickness in microns after phacoemulsification that was compared to preoperative values
Endothelial cell loss | Three months
  Corneal endothelial cell count (cell/ square mm) after phacoemulsification that was compared to preoperative values

SECONDARY OUTCOMES:
IOP | Three months
  Intraocular pressure in mmHg rise after after phacoemulsification

CONTACTS AND LOCATIONS:
Overall Officials: Khaled G Abueleinen, MD, PhD, Principal Investigator — Ophthalmology department, Faculty of Medicine Cairo University
Locations (1):
- Khaled G Abueleinen, Giza, Cairo Governorate, Egypt